CLINICAL TRIAL: NCT04056286
Title: Gastro-intestinal and Hormonal Responses to Systemic Inflammatory Disease: A Human Model Comprising Endotoxemia, Fast and Bed Rest.
Brief Title: Gastro-intestinal and Hormonal Responses to Systemic Inflammatory Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Food Ingrediens (Unknown); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Ketone Gastro study
Record Dates: First submitted 2019-07-29; First posted 2019-08-14 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-07

CONDITIONS: Motility Disorder; Catabolic State; Endotoxemia
Keywords: gastric emptying; gastro-intestinal motility; endotoxemia; catabolism; GLP-1; GIP
MeSH Terms: conditions — Endotoxemia | interventions — Whey

STUDY DESIGN:
Intervention Model Description: In a randomized crossover design, eight healthy lean young men will undergo either:
  i) Healthy conditions (overnight fast) + whey protein ii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest) + whey protein iii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest) + 3-OHB/whey protein
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessor will be blinded for all interventions and will recieve raw data sequentially numbered, and will therefore not know which data are from the same test object and which intervention was given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy + Whey (Experimental): Healthy (overnight fast)
  Interventions: Dietary Supplement: Whey
- Catabolic + Whey (Experimental): Catabolic (Inflammation (LPS) + 36 hour fast and bed rest)
  Interventions: Dietary Supplement: Whey
- Catabolic + 3-OHB / Whey (Experimental): Catabolic (Inflammation (LPS) + 36 hour fast and bed rest)
  Interventions: Dietary Supplement: 3-OHB/whey

INTERVENTIONS:
Dietary Supplement: Whey — 45 g whey protein + 20 g maltodextrin
  Arms: Catabolic + Whey; Healthy + Whey
Dietary Supplement: 3-OHB/whey — 50 g 3-OHB + 45 g whey protein + 20 g maltodextrin
  Arms: Catabolic + 3-OHB / Whey

SUMMARY:
The aim of this study is to describe hormonal responses and changes of the gastrointestinal (GI) tract during healthy and catabolic inflammatory conditions.

Participants will receive isocaloric, isonitrogenous beverages of either whey or 3-OHB+whey in a randomized crossover design during either healthy (overnight fast) or catabolic conditions (inflammation/endotoxemia + 36 h fast and bed rest).

DETAILED DESCRIPTION:
Background: Endotoxemia (LPS) is known to cause fever, inflammation and nausea, but the underlying mechanisms are unknown. In a human disease model comprising LPS-induced inflammation, 36 hour fast and bed rest the investigators want to investigate mechanisms accounting for the nausea and decreased food intake often observed in hospitalized patients.

Aim: This study aims to investigate total transit time and motility of the GI-tract together with the regulation of gut- and appetite hormones following catabolic conditions compared with healthy controlled conditions

Hypothesis:

Catabolic stress (endotoxemia/inflammation + 36 h fast and bed rest) induces GI-tract and hormonal changes compared with healthy conditions (overnight fast)

Interventions:

In a randomized crossover design, eight healthy, lean, young men will undergo either:

i) Healthy conditions (overnight fast) + whey protein

ii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest*) + whey protein

iii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest*) + 3-ketone/whey protein

Beverages will be isonitrogenous with 45 g whey protein + 20 g maltodextrin +/- 50 g of 3-OHB. Bolus/sip administration will be applied (1/3 bolus, 2/3 sip).Beverages will be isocaloric (fat will be added to interventions without 3-OHB)

*LPS will be administered (1 ng/kg) the day prior to the study together with fast and bed rest. On the study day LPS (0.5 ng/kg) will be injected.

ELIGIBILITY:
Inclusion Criteria:

* Between 20-40 years of age
* Body mass index between 20-30 kg/m^2
* Healthy
* Oral and written consent forms obtained prior to study day

Exclusion Criteria:

* Recent immobilization of an extremity that is not fully rehabilitated
* Lactose, lidocain or rubber allergies
* Current disease
* Use of anabolic steroids
* Smoking Former major abdominal surgery (Or current problems with the GI tract) >10 hours of exercise/weak Present ketogenic diets or high-protein diets Blood doner that does not want to discontinue blood donations until study completion Pending MR scan

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Difference in total gastro-intestinal transit time (healthy vs catabolic conditions) | Measured from intake of the Smartpill (together with the bolus of the protein beverages at t=210) until excretion with faeces (expected time frame: 2-5 days))
  Difference in total gastro-intestinal transit time measured by the Smartpill system between healthy and catabolic conditions. A pooled mean of the catabolic conditions will be used, if there is no difference between first and second exposure to LPS or "catabolic + whey" and "catabolic + 3-OHB/whey" interventions.

SECONDARY OUTCOMES:
Difference in gastric emptying (healthy vs catabolic conditions) | Measured from intake of the Smartpill (t = 210) until it leaves the ventricle (assessed by rise in pH levels, expected time frame: 2-7 hours)
  Difference in gastric emptying by Smartpill between healthy and catabolic conditions. A pooled mean of the two catabolic arms during the basal period will be represented
Difference in small intestine passage time (healthy vs catabolic conditions) | Measured from the timepoint where Smartpill leaves the ventricle until it enters the colon (assessed by specific predefined motility and pH patterns, expected timeframe 1-3 days)
  Difference in small intestine passage time by Smartpill between healthy and catabolic conditions. A pooled mean of the two catabolic arms during the basal period will be represented
Difference in colon passage time (healthy vs catabolic conditions) | Measured from the timepoint where Smartpill leaves the small intestine until it is excreted with faeces (assessed by specific predefined motility and pH patterns, expected timeframe 1-3 days)
  Difference in colon passage time by Smartpill between healthy and catabolic conditions. A pooled mean of the two catabolic arms during the basal period will be represented
Difference in GI motility (healthy vs catabolic conditions) | Measured from intake of the Smartpill (t = 210) until excretion with faeces (expected time frame: 2-5 days)
  Difference in GI motility measured by Smartpill pressure sensor between healthy and catabolic conditions. A pooled mean of the catabolic conditions will be used, if there is no difference between first and second exposure to LPS or "catabolic + whey" and "catabolic + 3-OHB/whey" interventions. A pooled mean of the two catabolic arms during the basal period will be represented
Difference in body temperature (healthy vs catabolic conditions) | Measured from intake of the Smartpill (t = 210) until excretion with faeces (expected time frame: 2-5 days)
  Difference in body temperature measured by Smartpill between healthy and catabolic conditions. A pooled mean of the two catabolic arms during the basal period will be represented
Difference in pH in the ventricle, small intestine and colon (healthy vs catabolic conditions) | Measured from intake of the Smartpill (t = 210) until excretion with faeces (expected time frame: 2-5 days)
  Difference in pH measured by Smartpill between healthy and catabolic conditions in the ventricle, small intestine and colon . A pooled mean of the catabolic conditions will be used, if there is no difference between first and second exposure to LPS or "catabolic + whey" and "catabolic + 3-OHB/whey" interventions. A pooled mean of the two catabolic arms during the basal period will be represented
Difference in gastric- and appetite hormones (GLP-1, GIP, PYY and ghrelin) (healthy vs catabolic conditions) | Measured at baseline and 30, 60, 90, 120 and 200 minutes after the beginning of the basal period
  Difference in hormones at baseline and throughout the basal period between healthy and catabolic conditions. A pooled mean of the two catabolic arms during the basal period will be represented
Difference in The Gastrointestinal Symptom Rating Scale (GSRS) (healthy vs catabolic conditions) | Given at timepoint t = 240 minutes
  Written assesment of various symptoms from the GI tract by a score from 0-6 (0 = no symptoms, 6 = very severe symptoms). A pooled mean of the two catabolic arms during the basal period will be represented
Difference in The Pain Catastrophizing Scale (PCS) (healthy vs catabolic conditions) | Given at timepoint t = 240 minutes
  Written assesment of pain-coping (score from 0-6 on each question, 0 = no worries, 6 = severe worrying). A pooled mean of the two catabolic arms during the basal period will be represented

CONTACTS AND LOCATIONS:
Overall Officials: Niels Moeller, Professor, Principal Investigator — Aarhus University Hospital and Institute of Clinical Medicine
Locations (1):
- Medical Reasearch labaratory, DoH, Aarhus University Hospital, Aarhus N, Danmark, Denmark